CLINICAL TRIAL: NCT07062276
Title: Analyze the Comparison of the Effectiveness of Kinesio ®and Dynamic Taping for De Quervain's Tenosynovitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID epidemic broke out shortly after the project started, and the number of cases coming to the hospital dropped sharply. Finally, the research project had to be terminated because it expired.
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-IJRB-N202111055
Record Dates: First submitted 2022-06-19; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2022-06

CONDITIONS: De Quervain's Tenosynovitis
Keywords: Kinesio ®; Dynamic taping; De Quervain's tenosynovitis
MeSH Terms: conditions — De Quervain Disease | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic taping (Experimental): The participants are taped by an occupational therapist trained in dynamic taping Level 1. Dynamic taping is to reduce the load on the extensor pollicis brevis (EPB) and abductor pollicis longus (APL) tendons and assist them to do motion. The patient's thumb metacarpophalangeal joint should be extended to the bottom, and the radiocarpal joint and thumb metacarpal carpal joint should be abducted to the bottom.Attach the starting end of the dynamic taping to the thumb, extend the patch to the length where the tension begins to be felt, and then attach it. The end end does not need to have tension on the forearm.
  Interventions: Other: Dynamic taping
- Kinesio (Active Comparator): The participants are taped by an occupational therapist who has received Class C training in kinesio. It provides sensory input and creates a subcutaneous space, thereby reaching the extensor pollicis brevis and abducting the pollicis longus. The relaxing and lifting pain relief effect. The length of the tape is measured from the interphalangeal joint through the metacarpal wrist joint to the distal radius of the case, and then the anchor point is under the interphalangeal joint, and then the extensor pollicis brevis, abductor pollicis longus stretch position, and the patch is along this Two muscles attach to the radius. The length of the second patch is about 2 to 3 grids. The middle of the patch is the anchor point, and the anchor point is at the tendon sheath (the place of pain). The two sides of the patch are pulled a little to create a subcutaneous space at the painful place to improve the pain condition.
  Interventions: Other: Kinesio ®

INTERVENTIONS:
Other: Dynamic taping — The dynamic tape is a new type of treatment. The material has high resilience. Its purpose is to help muscles and tissues absorb external forces and reduce tissue energy consumption.
  Arms: Dynamic taping
Other: Kinesio ® — Kinesio ®can effectively improve pain, edema, and assist functional movements. The elasticity of the patch creates wrinkles to relax the extensor pollicis brevis and the abductor longus muscle of the thumb.
  Arms: Kinesio

SUMMARY:
_De Quervain's tenosynovitis is inflammation and swelling of the tendon caused by repetitive thumb movements. In severe cases, the tendon sliding is limited, resulting in limited joint range of motion and affecting the quality of life. Kinesio ®can effectively improve pain, edema, and assist functional movements. The elasticity of the patch creates wrinkles to relax the extensor pollicis brevis and the abductor longus muscle of the thumb. The dynamic tape is a new type of treatment. The material has high resilience. Its purpose is to help muscles and tissues absorb external forces and reduce tissue energy consumption. By adjusting the human motor control mode, the work of injured tissues can be reduced, thereby improving the discomfort of sports injuries , accelerating the recovery of injured tissues and reducing the load of the extensor pollicis brevis tendon and the abductor pollicis longus tendon to assist the two tendons in their work. However, in the past, there was no dynamic taping applied to the study of De Quervain's tenosynovitis, and no dynamic taping and Kinesio ® applied to the study of De Quervain's tenosynovitis.

DETAILED DESCRIPTION:
PURPOSE:To explore the effectiveness of dynamic taping intervention in cases of stenosis of the De Quervain's tenosynovitis and the comparison with the effectiveness of Kinesio ®_ METHODS:The study collected data on cases of De Quervain's tenosynovitis in the rehabilitation department of a hospital in northern Taiwan. The tape was performed by a functional therapist trained Kinesio ® C level and dynamic tape level 1 course. The finger pinch strength and grip strength were assessed immediately before and after the intervention; The Patient-Rated Wrist Evaluation was used to assess pain and difficulty in performing activities of daily living. Obtain data after the case actually performs activities of daily living.

Data analysis: Nonparametric test will be used in the comparison of the pre- and post-evaluation data inter group. The analysis will be carried out using SPSS Statistic (v20.0) and α<0.05.

ELIGIBILITY:
Inclusion Criteria:

* An outpatient case of De Quervain's tenosynovitis referred by a rehabilitation physician.
* Symptoms need to last for more than 1 month.
* The case did not administer any medications and did not receive any rehabilitation treatment before being transferred to the occupational therapy department.
* The case will not have any uncomfortable reaction to Kinesio ® and dynamic taping.
* The case or the main caregiver can understand and cooperate with the relevant instructions of the research.
* Those who are willing to sign the consent form after fully understanding this research

Exclusion Criteria:

* Medical personnel have identified medical problems that may affect the test
* Authors of stroke recurrence or epilepsy during the intervention
* Participate in other experimental researches on rehabilitation efficacy during this research period
* Those who refuse to sign the subject's consent form

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Basic Demographic Information | Before the intervention.
  Questionnaires were used to collect gender, age, medical history, and duration of hand discomfort.
The Patient-Rated Wrist Evaluation(PRWE) | Change from Baseline and after intervention 24hours
  The 15-item self-assessment questionnaire is scored as an analogy score of 0-10. This assessment tool is divided into two categories for assessment and scored separately. The first category evaluates the pain status of the individual, with 0 being no pain at all and 10 being very severe pain; the second category assessing the difficulty in performing daily life, with 0 points In order to perform activities without difficulty, 10 points are difficult and cannot be performed
JAMAR® dynamometer | Change from Baseline and after intervention immediately
  To evaluate finger pinch strength and grip strength, the subjects were asked to use the maximum force to press the gripper for a total of 3 times. Each test required the subject to press for at least 5 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chou Chen, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellace JV, Healy D, Besser MP, Byron T, Hohman L. Validity of the Dexter Evaluation System's Jamar dynamometer attachment for assessment of hand grip strength in a normal population. J Hand Ther. 2000 Jan-Mar;13(1):46-51. doi: 10.1016/s0894-1130(00)80052-6. PMID 10718222
- [Background] Mostafavifar M, Wertz J, Borchers J. A systematic review of the effectiveness of kinesio taping for musculoskeletal injury. Phys Sportsmed. 2012 Nov;40(4):33-40. doi: 10.3810/psm.2012.11.1986. PMID 23306413
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] McNeill W, Pedersen C. Dynamic tape. Is it all about controlling load? J Bodyw Mov Ther. 2016 Jan;20(1):179-188. doi: 10.1016/j.jbmt.2015.12.009. Epub 2015 Dec 29. No abstract available. PMID 26891654
- [Background] Wolf JM, Sturdivant RX, Owens BD. Incidence of de Quervain's tenosynovitis in a young, active population. J Hand Surg Am. 2009 Jan;34(1):112-5. doi: 10.1016/j.jhsa.2008.08.020. Epub 2008 Dec 10. PMID 19081683